CLINICAL TRIAL: NCT00501280
Title: Biomarkers of Genetic Susceptibility in Environmentally-Exposed Migrant/Seasonal Farmworker Women and Their Children
Brief Title: Genetic Susceptibility in Migrant Farmworker Children
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2003-0350
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Epidemiology
Keywords: Epidemiology; Genetic Susceptibility; Migrant Farmworker Children; Migrant Education Program; Interview; Questionnaire
MeSH Terms: conditions — Genetic Predisposition to Disease | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 teaspoons of blood drawn and a urine sample from each mother/child.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MSF Women + their children: Blood and urine samples and interviews of Migrant or seasonal farmworker (MSF) woman + their children
  Interventions: Behavioral: Interview
- Non-MSF Women + their Children: Blood and urine samples and interviews of non-MSF women (women who have never worked in agriculture) and their children
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Interview by telephone or on-site in language of choice (English or Spanish), 60 to 70 minutes to complete the mother's and the child participants' questionnaires
  Other Names: Questionnaire

SUMMARY:
Primary Objectives:

1. To test the hypothesis that children whose mothers are Migrant/Seasonal Farmworkers (MSFs) (occupationally-exposed to pesticides) may be at a higher risk for exhibiting mutagen-induced DNA damage than children whose mothers and fathers are not MSFs.
2. To test the hypothesis that MSF mothers (occupationally-exposed to pesticides) may be at a higher risk for exhibiting mutagen-induced DNA damage than mothers who are not MSFs.

Secondary Objectives:

1. To test the hypothesis that both the extent of pesticide exposure and the type of polymorphisms in chemical detoxification genes and DNA repair genes contribute to the extent of cytogenetic damage found in children of MSF women.
2. To test the hypothesis that both the extent of pesticide exposure and the type of polymorphisms in chemical detoxification genes and DNA repair genes contribute to the extent of cytogenetic damage found in MSF mothers.
3. To test the hypothesis that the total concentration levels of organochlorine (OCP) and organophosphate (OP) pesticides will correlate with the mutagenic potency of the serum and urine of the children.
4. To test the hypothesis that the total concentration levels of OCP and OP pesticides will correlate with the mutagenic potency of the serum and urine of the mothers.
5. To test the hypothesis that inherited polymorphisms in the PON1 gene and its expression modulate the risk for OP genotoxicity measured by the inhibition of the acetylcholinesterase enzyme in MSF children.
6. To test the hypothesis that inherited polymorphisms in the PON1 gene and its expression modulate the risk for OP genotoxicity measured by the inhibition of the acetylcholinesterase enzyme in MSF mothers.

DETAILED DESCRIPTION:
Participants in this study are either MSF children and their mothers or non-MSF women (women who have never worked in agriculture) and their children. If a mother has more than one child in the school system, only one child can participate in the study. A major effort of this study is to collect, store and analyze blood and urine samples from MSF women children and a group of non-MSF women and children. Only the MSF children will be matched by ethnicity, sex, age (2 or more years), and place of residence to non-MSF children.

All mothers and children participants will be recruited from the school rosters of the Goose Creek Consolidated Independent School District in Harris County, and the La Joya School District in Hidalgo County. The names and addresses of all the children and their mothers are also included in the rosters. Each mother will be contacted by a telephone call or letter inviting her and her child to participate in the study. If they agree, they will then be asked if they would like to complete the interview by telephone with the interviewer from M. D. Anderson or prefer to do the interview at the on-site visit.

A bilingual interviewer will ask each child's mother if she and her child would like to participate in the study. The interviewer will ask each participating mother about her and her child's age, child's gender, her and her child's exposure to chemicals, medical history, places they have lived, places she has worked, family history of disease, reproductive and breast feeding histories, diet, alcohol and tobacco use. The interview will take from 60 to 70 minutes to complete the mother's and the child participants' questionnaires. All interviews will be completed by telephone or on-site in the language of choice (English or Spanish).

Two (2) members of the research team will collect the blood and urine samples, and transport them to M. D. Anderson since an overnight carrier is not available on the required days of collection. About 5 teaspoons of blood will be drawn and a urine sample will be collected. In addition, the height and weight of the mothers and the children will be measured. All blood and urine collected will be used only by the researchers involved in this study. If the child's mother agrees, the type(s) and levels of the pesticides detected will be provided to the child's physician for diagnostic purposes only. The data will be analyzed in a way that will help maintain confidentiality.

This is an investigational study. A total of 400 children participants and their mothers (N=400) will take part in this study. All 800 participants will be enrolled at UT MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Eligibility Criteria for the MSF Children: Children born of MSF women who are currently working in agriculture.
2. Enrolled in the Migrant Education Program
3. Ages 5-18, no gender restrictions
4. Residing in either Baytown (Harris County) or La Joya (Hidalgo County).
5. Eligibility Criteria for the non-MSF Children Population : Children attending the ESL Bilingual Education, Immigrant or Main Stream Programs in the same schools districts as the MSF Children
6. Whose mothers and/or fathers have never worked in agriculture.
7. Matched to the MSF children population by ethnicity, age plus/minus 2 years, gender, and residential status (i.e., MSF children in Baytown will be matched to non-MSF children from Baytown).
8. For MSF and non-MSF children: Children who have assented and whose mothers have signed the inform consent for participation in the study.
9. Eligibility criteria for MSF women: Women who have children 5-18 years of age who are currently enrolled in the Migrant Education Programs either in Baytown or La joya, TX, and who have conducted farmwork during the year of recruitment.
10. MSF women who have signed the inform consent for participation in the study.
11. Eligibility Criteria for Non-MSF women: Women who either themselves or their children's fathers have not performed farmwork, and whose 5-18 year old children (+/- 2 years) are enrolled in the ESL Bilingual, Immigrant or Main Stream Programs in the same school districts as the MSF children.
12. Non-MSF women who have signed an inform consent for participation in the study.

Exclusion Criteria:

1. Exclusion for the MSF children: Children who are not enrolled in the Migrant Education Program from either the Goose Creek Consolidated Independent School District, or the La Joya Consolidate School District.
2. Children who do not reside in Baytown or in La Joya, Texas.
3. Exclusion for the non-MSF children: Children who are not enrolled in the ESL Bilingual, Immigrant or Main Stream Programs from Baytown or La Joya, Texas.
4. Exclusion for both MSFs and non-MSF children: Children who have not assented or whose mothers have not signed the inform consent for study participation.
5. Exclusion for MSF women: Women whose children are not enrolled in the Migrant Education Program in Baytown or La Joya, Texas.
6. MSF women who do not reside either in Baytown or La Joya and who have not conducted farmwork during the year of recruitment.
7. MSF women who do not have children ages 5-18.
8. Exclusion for non-MSF women: Women whose children are not enrolled in either the Bilingual, Immigrant or Main Stream Programs in the school districts of Baytown or La joya, Tx.
9. Women who have not signed an informed consent for participation in the study.
10. Women who are not MSF but who do not have children ages 5-18 (+/- 2 years).

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Migrant or seasonal farmworker (MSF) woman who has a child attending the Migrant Education Program, or a child of a MSF woman, or a woman who has never worked in agriculture (non-MSF) but has a child attending the ESL Bilingual Education, Immigrant or the Main Stream Programs in the Goose Creek Consolidated School District in Harris County, TX, or in the La Joya School District in Hidalgo County, TX.
Sampling Method: Non-Probability Sample
Enrollment: 768 (Actual)
Dates: Start 2004-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
DNA damage [# of chromosome aberrations (CA)] calculated by exposure group | One time blood/urine collection from each mother/child

CONTACTS AND LOCATIONS:
Overall Officials: Maria A. Hernandez, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center official website — http://www.mdanderson.org